CLINICAL TRIAL: NCT02848755
Title: Neonatal Cranial Ultrasonography for Measuring Brain Volumes of Very Low Birth Weight Infants
Brief Title: Brain Volumes of Very Low Birth Weight Infants Measured by Cranial Ultrasonography
Status: Completed | Type: Observational
Sponsor: Zekai Tahir Burak Women's Health Research and Education Hospital (Other)
Collaborators: Netherlands: Ministry of Health, Welfare and Sports (Other Government)
Responsible Party: Principal Investigator, Gulsum Kadioğlu Simsek, Uzm Dr, Zekai Tahir Burak Women's Health Research and Education Hospital
Other Study IDs: 2016-Cr-USG-1
Record Dates: First submitted 2016-05-27; First posted 2016-07-28 (Estimated); Last update posted 2018-06-15 (Actual); Status verified 2018-06

CONDITIONS: Infant, Premature
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Cranial ultrasonography

SUMMARY:
Neonatal cranial ultrasound (US) remains the method of choice to detect brain injury in high risk preterm infants on neonatal intensive care units (NICU). It is a non-invasive, inexpensive bedside tool and examinations can be repeated as often as necessary without major disturbance of vulnerable infants. The anterior and posterior fontanelles from excellent acoustic windows to examine the deep midline and periventricular regions of the brain.Some data demonstrated that cerebral palsy can be accurately predicted with US. However, cranial US is not very suitable for investigating cortical regions or structures in the posterior fossa. There is limited data for very preterm infants.The investigators aimed to measure ventricular index, cranial height, biparietal diameter and calculate brain volume in a huge number of infants.

ELIGIBILITY:
Inclusion Criteria:

* both gender
* <1500 gr <32 week-
* 1-28 days neonates

Exclusion Criteria:

* Anomalies and no viability

Ages: 1 Day to 40 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All NICU preterm infants under 1500 gr
Sampling Method: Probability Sample
Enrollment: 341 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-05-09 (Actual); Study Completion 2018-06-09 (Actual)

PRIMARY OUTCOMES:
measurements of ventricular indexes of preterm infants | 12 months
  measuring distance with 2D USG
measurements of brain volumes of preterm infants | 12 months
  subtracting the ventricular volumes from the total brain volume measured with 2D

CONTACTS AND LOCATIONS:
Overall Officials: Fuat Emre Canpolat, Principal Investigator — Zekai Tahir Burak Hospital NICU
Locations (1):
- Zekai Tahir Burak NICU, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Rademaker KJ, Uiterwaal CS, Beek FJ, van Haastert IC, Lieftink AF, Groenendaal F, Grobbee DE, de Vries LS. Neonatal cranial ultrasound versus MRI and neurodevelopmental outcome at school age in children born preterm. Arch Dis Child Fetal Neonatal Ed. 2005 Nov;90(6):F489-93. doi: 10.1136/adc.2005.073908. Epub 2005 Jun 14. PMID 15956095
- [Derived] Isik S, Buyuktiryaki M, Simsek GK, Kutman HGK, Canpolat FE. Relationship between biparietal diameter/ventricular ratio and neurodevelopmental outcomes in non-handicapped very preterm infants. Childs Nerv Syst. 2021 Apr;37(4):1121-1126. doi: 10.1007/s00381-020-04960-5. Epub 2020 Nov 11. PMID 33175184
- [Derived] Simsek GK, Canpolat FE, Buyuktiryaki M, Okman E, Keser M, Ustunyurt Z, Kutman HGK. Developmental outcomes of very low birthweight infants with non-hemorrhagic ventricular dilatations and the relationships thereof with absolute brain volumes measured via two-dimensional ultrasonography. Childs Nerv Syst. 2020 Jun;36(6):1231-1237. doi: 10.1007/s00381-019-04464-x. Epub 2019 Dec 18. PMID 31853896